CLINICAL TRIAL: NCT05014451
Title: Pelvic Alignment in Relation to Standing Balance and Selective Motor Control in Children With Spastic Diplegia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Naglaa Ezzat Abd Allah Mahmoud, Teaching assistant, Cairo University
Other Study IDs: P.T.REC/012/003257
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy; Spastic Diplegia
Keywords: pelvic alignment; pelvic tilt, torsion, inclination; Formetric; Biodex; dynamic balance; selective motor control; SCALE
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be conducted to identify the relation between pelvic alignment and standing balance and also the relation between pelvic alignment and selective motor control in children with spastic diplegic cerebral palsy.

DETAILED DESCRIPTION:
In this study, pelvic alignment of children with diplegia will be evaluated using the Formetric instrument system. Their standing balance will be evaluated using the Biodex balance system, while selective voluntary motor control of lower extremities will be assessed using the Selective Control Assessment of the Lower Extremity scale (SCALE).

Results will be compared to find the correlation between pelvic alignment and standing balance and the correlation between pelvic alignment and selective motor control. Results can help clinicians to better address the problems of pelvic asymmetry in children with spastic diplegia to improve their overall balance and functional abilities.

ELIGIBILITY:
Forty children with spastic diplegia of both sexes will be selected with the following criteria:

Inclusion Criteria:

1. Their age will be ranged from 6 to 8 years.
2. The degree of their spasticity will be ranged from 1 to 1+ according to Modified Ashworth' Scale.
3. They will be on level Ⅰ or Ⅱ on Growth Motor Function Classification System (GMFCS).

Exclusion Criteria:

The Children will be excluded if they have one of the following:

1. Severe visual or hearing impairment.
2. Fixed deformities or surgical interventions in the lower extremities.
3. Botulinum toxin injections in the last 6 months.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with spastic diplegia, their height will not be less than 1 meter to meet the requirements of assessment by the Biodex and Formetric systems. They will be able to stand without the use of an assistive device and they will be able to follow instructions and understand given orders.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Pelvic alignment in relation to dynamic standing balance | 2 months
  Pelvic alignment will be assessed using the Formetric system, while standing balance will be assessed using the Biodex system then results will be compared to find the relation between pelvic alignment and dynamic standing balance in children with diplegia.
Pelvic alignment in relation to selective voluntary motor control of the lower extremities | 2 month
  Pelvic alignment will be assessed using the Formetric system, while selective motor control (SMC) of lower extremities will be assessed using Selective Control Assessment of the Lower Extremity scale (SCALE) then results will be compared to find the relation between pelvic alignment and selective motor control in children with diplegia.

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after completion of statistical analysis of the results.
Access Criteria: The data will be shared upon request.